CLINICAL TRIAL: NCT02830711
Title: The Impact of a 3-day High-altitude Mountain Trek on the Emotional States of Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, SHIH-HAO WANG, MD, Attending Physician, Chang Gung Memorial Hospital
Other Study IDs: 100-0921B
Record Dates: First submitted 2016-06-29; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Emotions
Keywords: happiness; anger; sadness; anticipation
MeSH Terms: interventions — Gene Expression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Other: Positive and Negative Affect Scale for Children — A 36-item instrument, including the Mood and Anxiety Symptom Questionnaire (MASQ)16 developed by Chang and Yeh and the Positive and Negative Affect Scale for Children developed by Watson and Clark

SUMMARY:
The mood was influenced by many factors in children. Sport, such as high-altitude mountain trek activity was thought benefit for human's mood and health. The expedition therapy was more and more popular in many schools recently. However, as the investigators best knowledge, there was no article discuss the relation between the mood and high-altitude mountain trek activity such as benefit influence in children. So, the investigators conduct the study.

Method: Demographic data will be recorded. The Professor Yeh's mood questionnaires were used to record the mood status of before and after the 3 days high-altitude mountain trek activity.

Statistical analyses: Participants rated their emotional states (happiness, sadness, anticipation, and anger) on a Likert scale. Each variable will be presented as descriptive statistics. Student t test or other suitable statistical method(s) will be used to determine the correction among the variables with scores of mood status. The paired t test or other suitable statistical method(s) will be used to determine the correction among the scores of mood status before and after the mountain activity. A difference was considered statistically significant if the p value were less than 0.05. All statistical analyses will be performed using SPPS statistical software for Windows, version 14 or more updated version.

ELIGIBILITY:
Inclusion Criteria:

* Sixth-grade elementary students who participated in a 3-day, 2-night high-altitude mountain walking trek from the trailhead (2,140 m above sea level) to the summit of Xue Mountain (3,886 m above sea level)
* Subject who provide the written informed consent from participants and their legal guardians before the distribution of the questionnaires.

Exclusion Criteria:

* Not Sixth-grade elementary students.
* Not finish the 3-day, 2-night high-altitude mountain walking trek from the trailhead (2,140 m above sea level) to the summit of Xue Mountain (3,886 m above sea level)
* Subject who do not provide the written informed consent from participants and their legal guardians before the distribution of the questionnaires.

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Sixth-grade elementary students who participated in a 3-day, 2-night high-altitude mountain walking trek from the trailhead (2,140 m above sea level) to the summit of Xue Mountain (3,886 m above sea level).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline Emotion States (happiness, anticipation, sadness, and anger) at 1 week after the trek. | 1 month before the trek and 1 week after the trek.
  A 36-item instrument, including the Mood and Anxiety Symptom Questionnaire was used to evaluate the four emotional states (happiness, anticipation, sadness, and anger). Specifically, 12 questions yielded the happy index, 10 questions yielded the sadness index, 9 questions yielded the anger index, and 5 questions yielded the anticipation index. A Likert scale ranging from 1 to 4 was used to evaluate individual items (1, strongly disagree; 2, disagree; 3, agree; and 4, strongly agree).

SECONDARY OUTCOMES:
Age | 1 month before the trek.
  Age in years
Gender | 1 month before the trek.
  Gender in male or female
Weight | 1 month before the trek.
  Weight in kilograms
Height | 1 month before the trek.
  Height in centimeters
Blood type | 1 month before the trek.
  Blood type in A, B, O, or AB blood types
Family configuration-father's and mother's Education level | 1 month before the trek.
  Junior high school, Senior high school, College, University, Graduate school, PH.D. or other
Family configuration-All Siblings | 1 month before the trek.
  1st, 2nd, 3rd, or 4th child
Family configuration-live with which family or families | 1 month before the trek.
  Live with both parents, mother only, father only, grandparents, or other relatives.

CONTACTS AND LOCATIONS:
Overall Officials: SHIH-HAO WANG, Principal Investigator — Chang Gung Memorial Hospital